CLINICAL TRIAL: NCT00136123
Title: Immediate Load of Dental Implants, Placed in Atrophic Upper and/or Lower Jaw of Partial or Complete Edentate Patients, According to Flapless Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/218
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implants (Experimental)
  Interventions: Procedure: Placement of functional loaded synthetic teeth after placement implants

INTERVENTIONS:
Procedure: Placement of functional loaded synthetic teeth after placement implants — Placement of functional loaded synthetic teeth after placement implants

SUMMARY:
This study will evaluate the placement of implants with minimal invasive techniques. Immediately after the placement of the implants, functional loaded synthetic teeth will be placed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Implant success at 0-3 years | At 0-3 years

SECONDARY OUTCOMES:
Prosthetic success | At the moment
Patient opinion | At same day

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be